CLINICAL TRIAL: NCT06809374
Title: Investigation of the Optimal Duration of Neoadjuvant Therapy for Resectable Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Kochi University (Other)
Responsible Party: Principal Investigator, Takehiro Okabayashi, Kochi Health Sciences Center, Kochi University
Other Study IDs: iON study
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Cancer Resectable
MeSH Terms: interventions — Gemcitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 100 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: gemcitabine — neoadjuvant therapy for resectable pancreatic cancer using gemcitabine +S1 or gemcitabine + nab-Paxitaxel

SUMMARY:
Investigating the Optimal Duration of Neoadjuvant Chemotherapy for Resectable Pancreatic Cancer to Determine the True Surgical Indication.

ELIGIBILITY:
Inclusion Criteria:

* radiologically resectable pancreatic cancer patients

Exclusion Criteria:

* a body weight loss of greater than 10% during the six months prior to surgery, the presence of distant metastases, or seriously impaired function of vital organs due to respiratory, renal, or heart disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: radiologically resectable pancreatic cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Investigating the Presence of Occult Metastatic Lesions Detected During Neoadjuvant Therapy. | within 6 months

IPD SHARING:
Plan to Share IPD: No